CLINICAL TRIAL: NCT02496104
Title: Habituation's Mechanisms in Preterm and Term Infants. Behavioral Evaluation: APIB (Assessment of Preterm Infant's Behavior). Assessment of the Cortical and Vegetative Responses
Brief Title: Habituation's Mechanisms in Preterm and Term Infants
Acronym: HABIPREMA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC14.0059
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Habituation, Psychophysiological; Preterm, Infant
Keywords: Preterm; Infant; Habituation; APIB
MeSH Terms: conditions — Substance-Related Disorders; Premature Birth | interventions — Sound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm infants: Preterm infants born between 25 weeks and 32 weeks + 6 days of gestation
  Interventions: Behavioral: Package n°1 of the APIB
- Term newborns: Infant born at term
  Interventions: Behavioral: Package n°1 of the APIB

INTERVENTIONS:
Behavioral: Package n°1 of the APIB
  Other Names: Sound and light stimulations

SUMMARY:
Each year in France, 7 % of newborns are born preterm (before 37 weeks of gestational age (GA)). The investigators called very preterm infants those who were born before 33 weeks of GA. These very preterm infants have a higher risk of developing neurological complications like developmental disabilities or cerebral palsy. To date, early assessment of these infants is difficult and not reliable enough to detect those who are at risks of developing neurological issues. Now, the investigators need to identify earlier these infants to provide them interventions to improve their development (physical therapy for example). Consequently, the investigators are examining a study whose aim is to assess preterm infants habituation. Habituation is the newborn ability to become familiar with new environmental stimulations (noise, light…). This habituation allows the newborn to maintain his sleep even at onset of a noise or light. To study this phenomenon in infants born preterm near to corrected term (around 40 weeks of postnatal GA), will allow us to better understand neurological development of these infants. The investigators plan to compare habituation skills of preterm infants near to their theorical date of birth (40 weeks of GA) to a population of infants born at term. The investigators will also study the link between habituation abilities and sleep quality as well as neurodevelopmental outcome at the corrected age of two years old.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants: preterm infants born from 25 weeks to 32 weeks + 6 days of gestation near to 36 weeks of gestation (corrected postnatal age)
* Term infants: term newborns with a gestational age between 39 and 41 weeks of gestation at day 3 with an Apgar ≥ 1 at 1 minute of life
* For both groups: normal neurological physical examination, written informed consent of the parents

Exclusion Criteria:

* no malformation or chromosomal abnormality, life threatening disease, administration of morphine or sedatives during the 24 hours before the study, context of maternal drug addiction, deafness, no psychoactive drug or anticonvulsivants during the last month of pregnancy for the term newborns, severe neurological disease

Ages: 2 Days to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants and term infants born in Brest University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-07-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the package n°1 of the APIB (Assessment of Premature Infant's Behaviour) | At 40 weeks of postnatal gestational age for the preterm infants and at 3 days old for the term newborns

SECONDARY OUTCOMES:
Salivary cortisol changes | Before and 30 minutes after the package n°1 of the APIB achievement
Oxy and deoxyhemoglobin changes in NIRS (Near-infrared Spectroscopy) | During APIB package n°1 fulfillment
Heart rate variations | During APIB package n°1 fulfillment
Oxymetry variations | During APIB package n°1 fulfillment
Brief Infant Sleep Questionnaire | At 6 and 12 months old (corrected age for the preterm infants)
Ages and Stages Questionnaire | At 24 months old (corrected age for the preterm infants)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel ROUE, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France